CLINICAL TRIAL: NCT04300920
Title: Prospective Treatment Efficacy in IPF Using Genotype for Nac Selection (PRECISIONS) Trial
Acronym: PRECISIONS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fernando J Martinez (Other)
Collaborators: University of Virginia (Other); University of Michigan (Other); Pulmonary Fibrosis Foundation (Other); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Three Lakes Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Fernando J Martinez, Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-12021232; 1U24HL145265-01A1 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Pulmonary Fibrosis; n-acetylcysteine; NAC
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 1:1 fashion to NAC or placebo, stratified by stable concomitant IPF therapy use (i.e., pirfenidone or nintedanib administered for at least 6 weeks prior to screening) versus no pirfenidone or nintedanib use. Participants will receive 600 mg NAC orally three times daily or matched placebo for 24 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and site personnel will not know which study treatment the participant is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine (Experimental): 600 mg oral N-acetylcysteine (NAC) three times daily for 24 months.
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Placebo tablet three times daily for 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — 600 mg N-acetylcysteine (NAC) oral tablets three times daily for 24 months.
  Other Names: NAC
  Arms: N-acetylcysteine
Drug: Placebo — Matching oral placebo tablet three times daily for 24 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of n-acetylcysteine (NAC) plus standard care with matched placebo plus standard of care in patients diagnosed with idiopathic pulmonary fibrosis (IPF) who have the TOLLIP rs3750920 TT genotype. The study will compare the time to a composite endpoint of relative decline in lung function [10% relative decline in forced vital capacity (FVC), first respiratory hospitalization, lung transplantation, or all-cause mortality]

The secondary objectives will be to examine the effect of NAC on the components of the primary composite endpoint, the rates of clinical events, change in physiology, change in health status, and change in respiratory symptoms.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled trial of NAC or placebo in about 200 participants with IPF with a TOLLIP rs3750920 TT genotype.

Eligible participants will be randomized in a 1:1 fashion to NAC or placebo, stratified by stable concomitant IPF therapy use (i.e., pirfenidone or nintedanib administered for at least 6 weeks prior to screening) versus no pirfenidone or nintedanib use. Participants will receive 600 mg NAC orally or matched placebo to take three times daily for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 years of age
* Diagnosed with IPF according to 2018 ATS/ERS/JRS/ALAT, confirmed by enrolling investigator
* Signed informed consent
* If taking pirfenidone or nintedanib, must be on stable dose for at least 6 weeks prior to enrollment visit
* Confirmed rs3570920 TT TOLLIP genotype

Exclusion Criteria:

* Pregnancy or planning to become pregnant
* Women of childbearing potential not willing to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year during study participation
* Significant medical, surgical or psychiatric illness that in the opinion of the investigator would affect subject safety, including liver and renal failure
* Receipt of an investigational drug or biological agent within the previous 4 weeks of the screening visit or 5 times the half-life, if longer
* Supplemental or prescribed NAC therapy within 60 days of enrollment
* Listed for lung transplantation at the time of screening
* History of lung cancer
* Inability to perform spirometry
* Forced vital capacity (FVC) less than 45% predicted, using the global lung function index (GLI) equation at Visit 1
* Active respiratory infection requiring treatment with antibiotics within 4 weeks of Visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Time to one of the following composite endpoint criteria: 10% relative decline in forced vital capacity (FVC), first respiratory hospitalization, lung transplant or death from any cause. | 24 months
  This is a composite endpoint of time to 10% relative decline in forced vital capacity (FVC), first respiratory hospitalization, lung transplant or death from any cause. Respiratory hospitalizations will be determined by a blinded clinical events classification (adjudication) committee.

SECONDARY OUTCOMES:
Time to one of the following composite criteria: 10% relative decline in FVC % predicted, first respiratory hospitalization, lung transplant or death from any cause. | 24 months
  This is a composite endpoint of time to 10% relative decline in FVC % predicted, based on the global lung initiative (GLI) reference equation, first respiratory hospitalization, lung transplant or death from any cause. Respiratory hospitalizations will be determined by a blinded clinical events classification (adjudication) committee.
Time to death from any cause | 24 months
Time to first respiratory hospitalization, lung transplant, or death from any cause | 24 months
  Respiratory hospitalizations will be determined by a blinded clinical events classification (adjudication) committee.
Time to 10% relative decline in FVC, lung transplant or death from any cause | 24 months
Time to lung transplant, or death from any cause | 24 months
Time to 10% relative decline in FVC %predicted, lung transplant, or death from any cause | 24 months
Time to first all-cause hospitalization, lung transplant, or death from any cause | 24 months
Annualized rate of respiratory hospitalizations | 24 months
Annualized rate of non-elective, all-cause hospitalizations | 24 months
Absolute change in FVC % predicted from randomization at 12 months | 12 months
Absolute change in FVC % predicted from randomization at 24 months | 24 months
Absolute change in FVC from randomization at 12 months | 12 months
Absolute change in FVC from randomization at 24 months | 24 months
Absolute change in diffusing capacity of the lung for carbon monoxide (DLCO) uncorrected for hemoglobin from randomization at 12 months | 12 months
Absolute change in DLCO uncorrected from randomization at 24 months | 24 months
Absolute change in patient reported outcomes scores for the Leicester Cough Questionnaire (LCQ) from randomization at 12 months. | 12 months
Absolute change in patient reported outcomes scores for the EuroQoL EQ-5D Questionnaire from randomization at 12 months. | 12 months
Change in patient reported outcomes scores for the University of California, San Diego Shortness of Breath (UCSD-SOB) Questionnaire from randomization at 12 months. | 12 months
Change in patient reported outcomes scores for the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire from randomization at 12 months. | 12 months
Change in patient reported outcomes scores for the St. George's Respiratory Questionnaire (SGRQ) from randomization at 12 months. | 12 months
Change in patient reported outcomes scores for the Leicester Cough Questionnaire (LCQ) from randomization at 24 months | 24 months
Change in patient reported outcomes scores for the EuroQoL EQ-5D Questionnaire from randomization at 24 months | 24 months
Change in patient reported outcomes scores for the University of California, San Diego Shortness of Breath (UCSD-SOB) Questionnaire from randomization at 24 months | 24 months
Change in patient reported outcomes scores for the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire from randomization at 24 months | 24 months
Change in patient reported outcomes scores for the St. George's Respiratory Questionnaire (SGRQ) from randomization at 24 months | 24 months
Proportion of participants with and number of treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation, and unanticipated problems | 24 months
Estimated time per six months free of 10% relative decline in FVC, first respiratory hospitalization, lung transplant or death from any cause. | 24 months
Estimated time per six months free of 10% relative decline in FVC % predicted, first respiratory hospitalization, lung transplant or death from any cause. | 24 months
Estimated time lived per six months (based on all-cause mortality). | 24 months
Average time per six months free of first respiratory hospitalization, lung transplantation or death from any cause. | 24 months
Average time per six months free of 10% relative decline in FVC, lung transplant, or death from any cause. | 24 months
Average time per six months free of lung transplant, or death from any cause. | 24 months
Average time per six months free of 10% relative decline in FVC % predicted, lung transplant, or death from any cause. | 24 months
Average time per six months free of all-cause hospitalization, lung transplant, or death from any cause. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, Principal Investigator — University of Massachusetts Chan Medical School; Imre Noth, MD, Principal Investigator — University of Virginia; Kevin Flaherty, MS, MD, Principal Investigator — University of Michigan; Cathie Spino, ScD, Principal Investigator — University of Michigan
Locations (25):
- United States (25):
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Piedmont Healthcare, Austell, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Lisa Lancaster, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The de-identified analytic data will be prepared as SAS transport files or ASCII comma-delimited files with accompanying codebooks that describe the data and data structure. The redaction will employ best practices and will be consistent with NHLBI data sharing policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after the end of the study or 2 years after the main paper reporting the results of the trial, whichever comes first.
Access Criteria: Data will be shared through the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC).
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Podolanczuk AJ, Kim JS, Cooper CB, Lasky JA, Murray S, Oldham JM, Raghu G, Flaherty KR, Spino C, Noth I, Martinez FJ; PRECISIONS Study Team. Design and rationale for the prospective treatment efficacy in IPF using genotype for NAC selection (PRECISIONS) clinical trial. BMC Pulm Med. 2022 Dec 13;22(1):475. doi: 10.1186/s12890-022-02281-8. PMID 36514019